CLINICAL TRIAL: NCT06061263
Title: The Patterns and Risk Factors of Relapse in Esophageal Squamous Cell Cancers Who Achieve Pathologic Complete Response to Neoadjuvant Chemoradiotherapy
Brief Title: Risk Factors of Relapse in Esophageal Squamous Cell Cancers Who Achieve PCR to Neoadjuvant Chemoradiotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianhua Fu, Professor, Sun Yat-sen University
Other Study IDs: 202212901
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: risk factor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCR patients with eaophageal squamous cell carcinomas: patients with esophageal squamous cell carcinoma (ESCC) patients who achieved pathologic complete response after neoadjuvant chemoradiotherapy (nCRT).
  Interventions: Other: follow up

INTERVENTIONS:
Other: follow up — collecttion of clinicopathological data from a prespectively collected databse, including survival data.

SUMMARY:
It has been reported that patients with esophageal squamous cell carcinoma who achieved pathological complete response (PCR) to neoadjuvant chemoradiotherapy have better survival than those with non-PCR. Howeve, there is still recurrent diseases developed in PCR patients after esophagectomy. Herein, we aimed to investgate the risk factors of recurrence in PCR patients.

DETAILED DESCRIPTION:
Between January 2008 and December 2018, a total of 96 patients with pathological complete response were enrolled in this study. Sterilized lymph nodes (SLN) were defined as those lymph nodes without residual tumor but with the presence of treatment response to neoadjuvant chemoradiotherapy. Prognostic factors for recurrence-free survival (RFS) were analyzed with univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

(1) patients with histopathologically confirmed ESCC;(2) patients received nCRT and radical esophagectomy in our hospital;(3) patients received the cisplabin plus or cisplain plus as the preoperative chemotherapy regimen; (4) those patients achieved PCR in the postoperative specimens (both primary tumor and resected lymph nodes).

Exclusion Criteria:

(1) patients who did not receive preoperative treatment or received preoperative chemotherapy alone;(2) patients who underwent Ivor-Lewis esophagectomy or Sweet esophagectomy;(3) patients who received preoperative chemotherapy other than NP or DP regimens;(4) patients with non-PCR to nCRT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all the ESCC patients with PCR to nCRT betwee 2008 and 2018 who received cisplabin plus or cisplain plus as the preoperative chemotherapy regimen.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 2008-2018
  recurrence-free survival (RFS) was calculated from the date of esophagectomy to the date of first detected recurrent disease

CONTACTS AND LOCATIONS:
Locations (1):
- Jianhua Fu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No